CLINICAL TRIAL: NCT04619446
Title: Dentoskeletal Changes of Twin Block Appliance and AdvanSync2 Appliance in Treatment of Skeletal Class II Malocclusion
Brief Title: Dentoskeletal Changes Produced by Growth Modification Appliances in Treatment of Skeletal Class II Malocclusion
Status: Completed | Type: Observational
Sponsor: Dr. Fareena Ghaffar (Other)
Responsible Party: Sponsor-Investigator, Dr. Fareena Ghaffar, Principal Investigator, Armed Forces Institute of Dentistry, Pakistan
Organization: Armed Forces Institute of Dentistry, Pakistan (Other)
Other Study IDs: AFIDPakistan
Record Dates: First submitted 2020-10-09; First posted 2020-11-06 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Class II Division 1 Malocclusion; Mandibular Retrognathism
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Removable Twin Block appliance group: Patient to be treated with removable twin block appliance that are known Class II skeletal and dental subjects.
  Interventions: Device: Removable Twin Block
- Fixed Functional Appliance AdvanSync group: Patients to be treated with fixed functional appliance, AdvanSync (Molar-to-Molar) Class II Corrector
  Interventions: Device: Fixed Functional , AdvanSync Appliance

INTERVENTIONS:
Device: Removable Twin Block — Twin block appliance (RFA) was introduced by William Clark in 1988. Many modifications for this appliance have been introduced lately. It has been named twin block for the characteristic of two unattached maxillary and mandibular plates with acrylic bite blocks, which makes 70o angle when come in contact with each other. Delta clasps are added for better retention of the appliance. This appliance plays a vital role in the treatment of mandibular retrognathia
  Groups: Removable Twin Block appliance group
Device: Fixed Functional , AdvanSync Appliance — AdvanSync2 (Ormco Co., Glendora, Calif) is a FFA being introduced recently as an advancement of Herbst appliance. It is a molar-to-molar appliance, connected by a telescopic rod, which allow for simultaneous treatment with braces. It is much smaller in size than the conventional Herbst appliance and reduces treatment duration up to six to nine months. It is much more acceptable by the patients as they complain less about sores and discomfort, and is esthetically pleasant since it's not visible in the mouth. Short arms of this appliance help to decrease irritation and discomfort of the patient, and helps to advance the mandible in a constant forward direction to encourage growth, and reduce malocclusion.
  Groups: Fixed Functional Appliance AdvanSync group

SUMMARY:
To compare dentoskeletal changes in patients with skeletal class II malocclusion induced due to treatment with orthodontic appliances; removable twin block appliance and fixed AdvanSync2 appliance in two different age group patients.

DETAILED DESCRIPTION:
41% of total orthodontic cases in Pakistani population are of class II malocclusion. Class II malocclusion is referred as maxillary protrusion, or mandibular retrusion, or combination of both, which can be corrected by treating the skeletal and dento-alveolar discrepancies. Out of many recommended treatment options, one can make use of either removable and/or fixed functional appliances. In the past, headgear has been used as a classic appliance for the correction of class II malocclusion. Other removable functional appliances (RFA) include Frankel, bionator and sander bite jumping appliances. Jasper jumper, Herbst appliance and mandibular protraction appliance (MPA) are the some of the fixed functional appliances (FFA) used. All these modalities are designed to modify the arches by re-orienting their position in both sagittal and vertical dimensions to bring about correction of main features of class II malocclusion.

AdvanSync2 (Ormco Co., Glendora, Calif) is a FFA being introduced recently as an advancement of Herbst appliance. It is a molar-to-molar appliance, connected by a telescopic rod, which allow for simultaneous treatment with braces. It is much smaller in size than the conventional Herbst appliance and reduces treatment duration up to six to nine months. It is much more acceptable by the patients as they complain less about sores and discomfort, and is esthetically pleasant since it's not visible in the mouth. Short arms of this appliance help to decrease irritation and discomfort of the patient, and helps to advance the mandible in a constant forward direction to encourage growth, and reduce malocclusion.

Twin block appliance (RFA) was introduced by William Clark in 1988. Many modifications for this appliance have been introduced lately. It has been named twin block for the characteristic of two unattached maxillary and mandibular plates with acrylic bite blocks, which makes 70o angle when come in contact with each other. This appliance is another treatment modality for cases with class II malocclusions, which can be carried out at an early age as well as the delayed treatment. However, delayed treatment was found to be much better for the patients in terms of less orthodontic visits.

AdvanSync2 appliance is a new treatment modality in orthodontics, and through thorough literature search, no study could be found in regard to this appliance in Pakistani population yet.Hence, the objective of this study was to compare dentoskeletal changes in skeletal class II malocclusion induced due to treatment with removable twin block appliance and fixed advanSync2 appliance in Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* Class II div 1 malocclusion with mandible being placed backwards (SNB angle <78o)
* Convex facial profile
* ANB angle to be >4 degree
* overall good oral health
* no previous orthodontic treatment being done
* peak of pubertal growth at the start of treatment

Exclusion Criteria:

* Subjects presenting with any developmental defects
* Asymmetrical facial profile
* Impacted / missing / supernumerary or transposed teeth

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A.F.I.D, Rawalpindi. Thirty patients ( 15 between cervical vertebral maturation (CVM) stage of 2-3 to be treated with removable functional applianc and remaining 15 between CVM stage of 4-5 to be treated with fixed functional appliance) with skeletal class II malocclusion, presented at the department of Armed forces institute of dentistry (AFID).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
effect of Class II malocclusion fixed functional bite corrector in comparison to class II removable bite corrector | 9 to 10 months
  efficacy of both the appliances is to be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Jan, Postgraduate, Study Director — Armed Forces institute of Dentistry (AFID)
Locations (1):
- Armed Forces Institute of Dentistry (AFID), Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No